CLINICAL TRIAL: NCT06792929
Title: The Effect of Virtual Reality Applications on Diagnostic Procedures Performed in Patients With Suspicious Thyroid Cancer
Brief Title: The Effect of Virtual Reality Applications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hamdiye ARDA SÜRÜCÜ, Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICLE-ARDASURUCU-003
Record Dates: First submitted 2025-01-18; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer; Virtual Reality Therapy; Ultrasound; Fine Needle Aspiration Biopsy; Thyroid Nodule (Diagnosis)
Keywords: Thyroid Cancer; Virtual Reality Therapy; Ultrasound; Thyroid Nodule; Fine needle aspiration biopsy
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Disease

STUDY DESIGN:
Intervention Model Description: virtual reality glasses group and control group
Who Masked: Participant
Masking Description: They do not know the experimental or control procedures that take place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality glasses group (Experimental): Patients will wear virtual reality glasses throughout the ultrasound-guided fine needle aspiration biopsy procedure.
  Interventions: Device: virtual reality glasses group
- Control group (No Intervention): patients without of virtual reality glasses

INTERVENTIONS:
Device: virtual reality glasses group — Patients will wear virtual reality glasses throughout the ultrasound-guided fine needle aspiration biopsy procedure.
  Arms: virtual reality glasses group

SUMMARY:
Thyroid nodules are a common health problem in the adult population. The majority of cancers are diagnosed by thyroid fine needle aspiration biopsy. Thyroid nodules generally show clinical findings in 1-5% of cases on physical examination and 20-70% on ultrasound examination. In diagnosis; Ultrasonography, fine needle aspiration biopsy, ultrasonography-guided fine needle aspiration biopsy, scintigraphy, computed tomography and magnetic resonance imaging are widely used. The fact that the thyroid fine needle aspiration biopsy procedure is painful, there is no speaking or coughing during the procedure, and in case of insufficient sample, the procedure must be performed several times. Its repetition causes fear and anxiety in patients. A combination of pharmacological and nonpharmacological methods for pain control likely provides the most effective pain relief for the patient. Distraction is one of the non-pharmacological methods used in pain control. Distraction is one of the most preferred methods to reduce pain in patients during diagnosis and treatment procedures. It is a method that allows patients to control and reduce the symptoms they experience by focusing their attention on a different point.The aim of this study is to examine the effect of using a motivational video with virtual reality glasses to distract attention during the biopsy procedure on pain, stress and fear in individuals with suspected thyroid cancer.

DETAILED DESCRIPTION:
Research Type:

It was designed as a randomized controlled experimental study.

Research Population and Sample:

The research sample will consist of patients with suspected thyroid mass who applied to a University Hospitals. The sample of the research is aimed to be 100 volunteer diabetic patients who applied to the University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected thyroid mass
* No dizziness problem
* No vision problems

Exclusion Criteria:

* Mental health problems that may prevent wearing virtual reality glasses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before and immediately after ultrasound guided fine needle aspiration biopsy procedure
  The scale is used to assess subjectively perceived pain. It is a 10 cm (100 mm) ruler with no pain on one end and the "most severe pain" on the other. The individuals participating in the study are asked to mark the intensity of pain they are currently feeling, explaining that the number "0" on the scale means "I feel no pain" and that the intensity of pain increases as the numbers increase, and the number "10" means "I feel the most severe pain". An increase in the score obtained from the scale in the assessment indicates that the pain is increasing. Each patient will be administered two times.

SECONDARY OUTCOMES:
Fear of Pain Scale-III | Before and immediately after ultrasound guided fine needle aspiration biopsy procedure
  Fear of Pain Scale-III is a 30-item, 5-point Likert type scale developed to measure fear and/or anxiety about pain. The scale consists of 3 sub-dimensions and there are 10 items in each dimension. Scale items for fear of severe pain are 1, 3, 5, 6, 9, 10, 13, 18, 25, 27; scale items for fear of mild pain 2, 4, 7, 12, 19, 22, 23, 24, 28, 30; The scale items for fear of medical pain are 8, 11, 14, 15, 16, 17, 20, 21, 26, 29. In evaluating the score of the scale, which has no inverse expression, the items are rated with a Likert-type scoring ranging from 1 to 5 (1- never, 2-a little, 3-quite a bit, 4-a lot, 5-extremely). 1-refers to never feeling fear, 5-expresses excessive fear. The lowest possible score in total is 30 and the highest score is 150. The lowest score that can be obtained for the sub-dimensions is 10 and the highest score is 50. A high score on the scale indicates that the individual's fear of pain is also high.
Beck Anxiety Scale | Before and immediately after ultrasound guided fine needle aspiration biopsy procedure
  It measures the severity of anxiety symptoms experienced by individuals. Consisting of 21 items, scored between 0-3; It is a scale filled by the patient himself. Score Range is 0-63. Anxiety levels of the patients according to the scores obtained; 0-7 points are classified as no anxiety, 8-15 points as mild anxiety, 16-25 points as moderate anxiety, and 26 and above points as severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle Univertsity, Diyarbakır, South East, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No